CLINICAL TRIAL: NCT02884440
Title: Transverse Abdominis Plane Block for Anterior Approach Spine Surgery: A Prospective Randomized Study
Brief Title: Transverse Abdominis Plane Block for Anterior Approach Spine Surgery
Acronym: TAP ALIF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 35RC15_8933_TAP-ALIF
Record Dates: First submitted 2016-08-22; First posted 2016-08-31 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Spine Surgery; Low Back Pain; Spondylolisthesis
MeSH Terms: conditions — Low Back Pain; Spondylolisthesis | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP block ropivacaine (Experimental): Bilateral ultrasound guided with 15 ml ropivacaine 5mg/ml on each side under general anesthesia at the end of the intervention
  Interventions: Drug: TAP block ropivacaine; Drug: General anesthesia
- TAP block placebo (Placebo Comparator): Bilateral ultrasound guided with 15 ml saline on each side under general anesthesia at the end of the intervention
  Interventions: Drug: TAP block placebo; Drug: General anesthesia

INTERVENTIONS:
Drug: TAP block ropivacaine
  Arms: TAP block ropivacaine
Drug: TAP block placebo
  Arms: TAP block placebo
Drug: General anesthesia — Induction PROPOFOL 10mg/ml REMIFENTANIL 50 μg/ml CISATRACURIUM 2mg/ml if necessary DEXAMETHASONE 8 mg KETAMINE 0,15mg/kg Maintenance PROPOFOL 10mg/ml REMIFENTANIL 50 μg/ml

SUMMARY:
Therapeutic, prospective, randomized, double blind, placebo-controlled, in intention to treat, monocentric study to evaluate the analgesic efficacy of a bilateral TAP block after spine surgery with 24 hours morphine consumption

DETAILED DESCRIPTION:
ALIF is a commonly performed procedure for the treatment of degenerative diseases of the lumbar spine or spondylolisthesis. This technique has many advantages attributed to the absence of posterior spinal muscular pain, a more direct visualization of the disk space, lower incidence of neurological injuries… However, patients experienced moderate to high post operative parietal abdominal pain due to this specific anterior approach. The systematic need for opioids administration may cause many complications and delay the post operative recovery time. The TAP block has been described as an effective pain control technique after various lower abdominal surgeries, reducing both pain scores and 24 hours opioids consumption. However the analgesic efficacy of this technique on specific parietal abdominal pain experienced after spine surgery by anterior approach is not clear

ELIGIBILITY:
Inclusion Criteria:

* Patient with age above 18 years old
* Patients scheduled for spine surgery by anterior approach
* Patient who signed an informed consent form

Exclusion Criteria:

* Allergy to ropivacaine
* Weight < 50 kg
* Contra indication to TAP block : sepsis in the point of draining, bleeding disorder
* Contra indication to paracetamol: severe hepatic insufficiency
* Contra indication to ketoprofen: age ≥ 75 years, renal insufficiency, previous gastric ulcer, allergy
* Contra indication to nefopam: severe cardiac insufficiency, glaucoma, prostate hypertrophy, allergy
* Known allergy to active substance or at least to one excipient (propofol, paracetamol, morphine, remifentanil, cisatracurium)
* Allergy to fentanyl, atracurium, or benzin sulfonic acid derivative, to propacetamol
* Convulsions or previous convulsive disorder
* Severe respiratory insufficiency
* Abnormal hemostasis or anticoagulant treatment because of possible intramuscular injection
* Morphine intake 24 hours before surgery
* Chronic use of morphine, gabapentin, pregabalin
* Pregnancy or breastfeeding
* Patient unable to use Patient Controlled Analgesia (PCA) (old patient depends…)
* Patients subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
Morphine consumption in the first 24 hours after spine surgery by anterior approach | 24 hours

SECONDARY OUTCOMES:
Morphine consumption in the first 48 hours after spine surgery by anterior approach | 48 hours
Assessment of pain | 1, 6, 12, 24 and 48 hours
  Numerical Analogue score
Assessment of post operative nausea or vomiting | 48 hours
  Occurence of nausea or vomiting episodes over 48 hours
Delay before first morphine administration | Day 1
  Number of hours between end of surgery and first morphine administration
Delay before the first lift | Day 1
  Number of hours between end of surgery and the first lift
Delay before resumption of transit | Day 1
  Number of days between end of surgery and resumption of transit
Duration of hospitalization | Day 1
Patient satisfaction | 48 hours
  Satisfaction questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coquet A, Sion A, Bourgoin A, Ropars M, Beloeil H. Transversus abdominis plane block for anterior lumbar interbody fusion: a randomized controlled trial. Spine J. 2023 Aug;23(8):1137-1143. doi: 10.1016/j.spinee.2023.03.013. Epub 2023 Apr 7. PMID 37031893